CLINICAL TRIAL: NCT04378114
Title: Impact of Acetaminophen on Performance of Guardian™ Sensor (3) in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: CIP333
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Results first posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Subjects with diabetes wearing Guardian™ Sensor (3). C algorithm applied retrospectively (Experimental): Subjects wear Guardian™ Sensor (3) over 7 days and undergo one frequent sample test (FST). C sensor algorithm applied retrospectively to raw sensor data.
  Interventions: Device: Guardian™ Sensor (3) connected to a Guardian™ Connect Transmitter. C sensor algorithm applied retrospectively to raw sensor data.; Drug: Acetominophen
- Subjects with diabetes wearing Guardian™ Sensor (3). Zeus algorithm applied retrospectively (Experimental): Subjects wear Guardian™ Sensor (3) over 7 days and undergo one FST. Zeus sensor algorithm applied retrospectively to raw sensor data.
  Interventions: Device: Guardian™ Sensor (3) connected to a Guardian™ Connect Transmitter. Zeus sensor algorithm applied retrospectively to raw sensor data.; Drug: Acetominophen

INTERVENTIONS:
Device: Guardian™ Sensor (3) connected to a Guardian™ Connect Transmitter. C sensor algorithm applied retrospectively to raw sensor data. — Characterize the impact of acetaminophen ingestion on the accuracy of Guardian™ Sensor (3) when C sensor algorithm is used.
  Arms: Subjects with diabetes wearing Guardian™ Sensor (3). C algorithm applied retrospectively
Device: Guardian™ Sensor (3) connected to a Guardian™ Connect Transmitter. Zeus sensor algorithm applied retrospectively to raw sensor data. — Characterize the impact of acetaminophen ingestion on the accuracy of Guardian™ Sensor (3) when Zeus sensor algorithm is used.
  Arms: Subjects with diabetes wearing Guardian™ Sensor (3). Zeus algorithm applied retrospectively
Drug: Acetominophen — One time administration of acetaminophen.

SUMMARY:
The purpose of this study is to characterize the impact of acetaminophen ingestion on the performance of the Guardian™ Sensor (3) (i.e., C algorithm and Zeus algorithm) in subjects age 18 - 80 years.

DETAILED DESCRIPTION:
The study is a multi-center, prospective, study without controls. The purpose of this study is to characterize the impact of acetaminophen ingestion on the performance of the Guardian™ Sensor (3) (i.e., C algorithm and Zeus algorithm) in subjects age 18 - 80 years.

ELIGIBILITY:
Inclusion Criteria:

1. Individual is 18 - 80 years of age at time of enrollment.
2. Subject has a clinical diagnosis of type 1 or type 2 diabetes for a minimum of 6 months duration as determined via medical record/ source documentation by an individual qualified to make a medical diagnosis.
3. Subject has adequate venous access as assessed by investigator or appropriate staff.

Exclusion Criteria:

1. Subject has history of allergy to acetaminophen or has been told by a health care provider they may not ingest acetaminophen
2. Subject reports history of liver cirrhosis or liver problems that a health care provider told them they should not use acetaminophen because of liver disorder.
3. Subject will not tolerate tape adhesive in the area of Guardian™ Sensor (3) placement as assessed by a qualified individual.
4. Subject has any unresolved adverse skin condition in the area of sensor or device placement (e.g., psoriasis, rash, Staphylococcus infection).
5. Subject is actively participating in an investigational study (e.g., drug or device) wherein he/she has received treatment from an investigational study (drug or device) in the last 2 weeks prior to Visit 1. (Please note participation in an observational study is acceptable.)
6. Subject is female of child-bearing potential and has a pregnancy screening test that is positive.
7. Subject is female of child-bearing potential and who is sexually active should be excluded if she is not using a form of contraception deemed reliable by investigator.
8. Subject is female and plans to become pregnant during the course of the study.
9. Subject is breast feeding.
10. Subject has a chronic heavy alcohol use as determined by investigator.
11. Subject has a history of a seizure disorder.
12. Subject has a hematocrit (Hct) more than 10% below the lower limit of normal reference range (please note that patients may use prior blood draw from routine care as long as done within 6 months of screening and report of lab placed with subject source documents).
13. Subject has a history of adrenal insufficiency.
14. Subject is a member of the research staff involved with the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2020-07-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - AMCR Institue, Escondido, California
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - Diablo Clinical Research, Walnut Creek, California
  - Barbara Davis Center - Adults, Aurora, Colorado
  - "Atlanta Diabetes Associates, Atlanta, Georgia
  - Rainier Clinical Research Center, Inc., Renton, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 104 subjects consented and enrolled in the overall study. Of them, 102 subjects were eligible.
Groups:
- Subjects With Diabetes Wearing Guardian™ Sensor (3): Subjects wearing two Guardian™ Sensor (3) on the arm and abdomen over 7 days and undergoing one Frequent Sample Testing (FST).
  One time acetaminophen (1000 mg) ingestion was administered while wearing Guardian™ Sensor (3) connected to a Guardian™ Connect Transmitter. The impact of acetaminophen ingestion on the accuracy of Guardian™ Sensor (3) using Zeus and C Algorithm was characterized.
Period: Overall Study
Arm/Group | Subjects With Diabetes Wearing Guardian™ Sensor (3)
Started | 102
Completed | 97
Not Completed | 5
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Arm/Group | Subjects With Diabetes Wearing Guardian™ Sensor (3)
Number analyzed (Participants) | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19
  Not Hispanic or Latino | 83
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 102

OUTCOME MEASURES:

1. Primary Outcome: Bias (mg/dL) Between the Guardian™ Sensor (3) Values and Yellow Springs Instrument™ (YSI™) Plasma Glucose
Description: Bias (mg/dL) between the Guardian™ Sensor (3) values and YSI™ plasma glucose values 1 hour before through 5 hours after ingestion of acetaminophen; results are reported hourly.
  Bias = Mean of [Guardian™ Sensor (3) values - YSI™ plasma glucose values].
Time Frame: Frequent sample testing recordings from the 6-hour period leading to and after Acetaminophen ingestion on day 4 or day 5 reported
Population: Subjects with at least 1 sensor-YSI paired point during the 1 hour before and 5 hours after ingestion of acetaminophen
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Subjects With Diabetes Wearing Guardian™ Sensor (3), Zeus Algorithm, Arm: Subjects wearing Guardian™ Sensor (3) on the arm over 7 days and undergoing one Frequent Sample Testing (FST).
  One time acetaminophen (1000 mg) ingestion was administered while wearing Guardian™ Sensor (3) connected to a Guardian™ Connect Transmitter. The impact of acetaminophen ingestion on the accuracy of Guardian™ Sensor (3) using Zeus Algorithm was characterized.
- Subjects With Diabetes Wearing Guardian™ Sensor (3), Zeus Algorithm, Abdomen: Subjects wearing Guardian™ Sensor (3) on the abdomen over 7 days and undergoing one Frequent Sample Testing (FST).
  One time acetaminophen (1000 mg) ingestion was administered while wearing Guardian™ Sensor (3) connected to a Guardian™ Connect Transmitter. The impact of acetaminophen ingestion on the accuracy of Guardian™ Sensor (3) using Zeus Algorithm was characterized.
- Subjects With Diabetes Wearing Guardian™ Sensor (3), C Algorithm, Arm: Subjects wearing Guardian™ Sensor (3) on the arm over 7 days and undergoing one Frequent Sample Testing (FST).
  One time acetaminophen (1000 mg) ingestion was administered while wearing Guardian™ Sensor (3) connected to a Guardian™ Connect Transmitter. The impact of acetaminophen ingestion on the accuracy of Guardian™ Sensor (3) using C Algorithm was characterized.
- Subjects With Diabetes Wearing Guardian™ Sensor (3), C Algorithm, Abdomen: Subjects wearing Guardian™ Sensor (3) on the abdomen over 7 days and undergoing one Frequent Sample Testing (FST).
  One time acetaminophen (1000 mg) ingestion was administered while wearing Guardian™ Sensor (3) connected to a Guardian™ Connect Transmitter. The impact of acetaminophen ingestion on the accuracy of Guardian™ Sensor (3) using C Algorithm was characterized.
Arm/Group | Subjects With Diabetes Wearing Guardian™ Sensor (3), Zeus Algorithm, Arm | Subjects With Diabetes Wearing Guardian™ Sensor (3), Zeus Algorithm, Abdomen | Subjects With Diabetes Wearing Guardian™ Sensor (3), C Algorithm, Arm | Subjects With Diabetes Wearing Guardian™ Sensor (3), C Algorithm, Abdomen
Number analyzed (Participants) | 102 | 102 | 102 | 102
mg/dL
  (-1,0] hour | -0.46 (16.05) | 0.86 (15.71) | -4.78 (9.79) | -4.45 (12.22)
  (0,1] hour | 14.83 (20.23) | 19.57 (19.35) | 10.64 (14.89) | 13.28 (19.56)
  (1,2] hour | 25.42 (18.74) | 29.92 (19.90) | 18.86 (15.19) | 21.99 (21.27)
  (2,3] hour | 19.60 (16.74) | 21.85 (15.31) | 13.52 (12.26) | 14.52 (15.31)
  (3,4] hour | 14.70 (15.29) | 17.22 (14.33) | 8.77 (12.36) | 8.98 (12.95)
  (4,5] hour | 11.12 (14.81) | 13.40 (13.80) | 4.93 (12.49) | 4.35 (13.70)

2. Secondary Outcome: Mean Absolute Relative Difference (MARD, %) Between the Guardian™ Sensor (3) Values and YSI™ Plasma Glucose
Description: Mean absolute relative difference (MARD, %) between the Guardian™ Sensor (3) values and YSI™ plasma glucose 1 hour before through 5 hours after ingestion of acetaminophen; results are reported hourly.
  Mean Absolute Relative Difference = Mean of ([absolute difference of Guardian™ Sensor (3) values and YSI™ plasma glucose / YSI™ plasma glucose] * 100%).
Time Frame: as for outcome 1
Population: Subjects with at least 1 sensor-YSI paired point during the 1 hour before and 5 hours after ingestion of acetaminophen
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Subjects With Diabetes Wearing Guardian™ Sensor (3), Zeus Algorithm, Arm | Subjects With Diabetes Wearing Guardian™ Sensor (3), Zeus Algorithm, Abdomen | Subjects With Diabetes Wearing Guardian™ Sensor (3), C Algorithm, Arm | Subjects With Diabetes Wearing Guardian™ Sensor (3), C Algorithm, Abdomen
Number analyzed (Participants) | 102 | 102 | 102 | 102
Percent
  (-1, 0] hour | 8.45 (6.52) | 8.38 (7.37) | 5.99 (4.24) | 6.56 (4.92)
  (0, 1] hour | 16.65 (10.72) | 18.02 (12.41) | 13.22 (8.17) | 16.09 (9.92)
  (1, 2] hour | 21.26 (15.16) | 24.22 (15.73) | 15.83 (12.89) | 18.60 (15.02)
  (2, 3] hour | 17.72 (12.95) | 18.44 (12.12) | 12.24 (9.40) | 12.92 (10.16)
  (3, 4] hour | 15.58 (11.16) | 15.87 (11.78) | 9.60 (7.28) | 10.06 (7.92)
  (4, 5] hour | 13.98 (10.48) | 13.87 (11.53) | 8.52 (6.12) | 8.70 (7.72)

3. Secondary Outcome: Percentage of Guardian™ Sensor (3) Values That Were Within 20% of YSI™ Plasma Glucose Values
Description: Percentage of Guardian™ Sensor (3) values within 20% of YSI™ plasma glucose value (±20 mg/dL [1.1 mmol/L] when YSI™ value less than or equal to (≤) 80 mg/dL [4.4 mmol/L]) during the 1 hour before through 5 hours after ingestion of acetaminophen; results are reported hourly.
  20% agreement = Number of Guardian™ Sensor (3) values within 20% (±20 mg/dL) of YSI™ plasma glucose value / Total number of paired Guardian™ Sensor (3) and YSI™ plasma glucose points * 100%.
Time Frame: as for outcome 1
Population: Subjects with at least 1 sensor-YSI paired point during the 1 hour before and 5 hours after ingestion of acetaminophen
Measure: Mean (Standard Deviation); unit: Percentage of readings
Arm/Group | Subjects With Diabetes Wearing Guardian™ Sensor (3), Zeus Algorithm, Arm | Subjects With Diabetes Wearing Guardian™ Sensor (3), Zeus Algorithm, Abdomen | Subjects With Diabetes Wearing Guardian™ Sensor (3), C Algorithm, Arm | Subjects With Diabetes Wearing Guardian™ Sensor (3), C Algorithm, Abdomen
Number analyzed (Participants) | 102 | 102 | 102 | 102
Percentage of readings
  (-1, 0] hour | 93.27 (21.36) | 94.44 (21.49) | 99.03 (5.33) | 96.40 (16.29)
  (0, 1] hour | 68.90 (29.84) | 67.82 (27.45) | 77.97 (20.64) | 73.70 (25.44)
  (1, 2] hour | 54.82 (44.92) | 47.37 (42.56) | 72.08 (39.05) | 65.43 (42.64)
  (2, 3] hour | 66.57 (43.87) | 64.64 (45.14) | 78.92 (36.93) | 78.91 (35.92)
  (3, 4] hour | 73.05 (40.85) | 73.91 (41.88) | 88.27 (25.64) | 87.97 (27.98)
  (4, 5] hour | 76.88 (40.13) | 75.97 (40.11) | 93.44 (17.67) | 91.03 (24.17)

ADVERSE EVENTS:
Time Frame: Throughout the course of the study, with an average of 25 days
Arm/Group | Subjects With Diabetes Wearing Guardian™ Sensor (3)
All-Cause Mortality (participants affected / at risk) | 0/102
Serious Adverse Events (participants affected / at risk) | 0/102
Other Adverse Events (participants affected / at risk) | 6/102
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects With Diabetes Wearing Guardian™ Sensor (3) (N=102)
Infusion site pruritus (Gastrointestinal disorders) | 1 (1)
Medical device site erythema (General disorders) | 2 (2)
Medical device site haemorrhage (General disorders) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/14/NCT04378114/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-13): https://cdn.clinicaltrials.gov/large-docs/14/NCT04378114/SAP_001.pdf